CLINICAL TRIAL: NCT07147959
Title: PET-Based Imaging to Evaluate the Distribution of Radiolabeled CIT-013 in Patients With Inflammatory Mediated Immune Disease
Brief Title: PET-Based Imaging of Radiolabeled CIT-013
Acronym: Cityview
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Citryll BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CITRYLL004
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: RA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [89Zr]Zr-CIT-013 (Experimental)
  Interventions: Drug: [89Zr]Zr-CIT

INTERVENTIONS:
Drug: [89Zr]Zr-CIT — radiolabelled CIT-013

SUMMARY:
Inflammatory mediated immune diseases (IMIDs), such as rheumatoid arthritis (RA) and hidradenitis suppurativa (HS), are characterized by chronic inflammation resulting from an aberrant immune response. Recent studies have identified neutrophil extracellular traps (NETs) as key contributors to the pathology of these diseases. CIT-013 is a novel humanized monoclonal antibody designed to inhibit NET release and enhance phagocytosis, offering a new potential therapeutic strategy for RA and HS. Previous clinical trials have demonstrated that CIT-013 is well tolerated in both healthy volunteers and patients with RA, with evidence of reduced NET formation and positive effects in active RA cases. Since NET-related inflammation primarily occurs in local tissues, understanding CIT-013's distribution beyond blood measurements is crucial for evaluating its therapeutic potential. This trial therefore uses radiolabeled CIT-013 and Positron Emission Tomography-Computed Tomography (PET-CT) imaging, along with lymph node biopsies, to evaluate the distribution of CIT-013 and target engagement in patients with IMIDs.

ELIGIBILITY:
Inclusion Criteria:

* Female (of non-childbearing potential) or male between 60-85 years of age (both inclusive).
* For male participants with female partners of child-bearing potential, an adequate form of contraception must be adhered to, and men must refrain from donating sperm, prior to entry into the trial and for a further 6 months after IP administration.
* Willing and able to provide written, informed consent.

Exclusion Criteria:

* Diagnosed with RA according to the 2010 classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) ≥ 6 months prior to screening (diagnosis based on medical records).

Participants in Cohort A (active RA) must furthermore meet the following criteria:

- Disease Activity Score 28 (DAS28) C-Reactive Protein (CRP) (DAS28-CRP) ≥ 4.2 AND ≥ 1 Swollen Joint AND ≥ 1 Tender Joint prior to screening.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of radiolabeled CIT-013 in patients with IMIDs | 24 hours
  Whole body PET-CT imaging 24 hours (D2) after IP administration. In addition to visual assessment, uptake of [89Zr]-DFO-CIT013 will be quantified per organ(-system). In vivo distribution profiles will be evaluated per cohort to determine ranges of uptake per organ(-system) and between cohorts to compare uptake in different IMIDs

SECONDARY OUTCOMES:
safety and tolerability of CIT-013 in patients with IMIDs. | Day 29
  Frequency and severity of treatment-emergent adverse events (TEAE) throughout the trial period, including clinically relevant findings and ADAs.

CONTACTS AND LOCATIONS:
Locations (1):
- NL-01, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided